CLINICAL TRIAL: NCT00122148
Title: Can Vignettes be Used to Improve Practice and Outcomes?
Brief Title: Can Vignettes Be Used to Improve Practice & Outcome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Jain, Sharad - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: IIR 01-189
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2006-08

CONDITIONS: Healthy
Keywords: Quality of health care; Feedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Behavioral: Feedback on provision of care

INTERVENTIONS:
Behavioral: Feedback on provision of care

SUMMARY:
This is a pilot study to first measure the cross-sectional relationship between variations in physicians� vignette scores and aggregated scores of individual physicians� patient health outcomes; and second to (longitudinally) determine whether feedback of vignette scores improves physicians� clinical performance as measured by vignettes

DETAILED DESCRIPTION:
1. Study Design: Physicians will complete computerized vignettes for four conditions � diabetes, coronary artery diseases (CAD), chronic obstructive pulmonary disease (COPD), and depression. We will collect retrospective outcomes data and develop composite outcome measures for on two conditions, Diabetes and CAD. For the longitudinal analysis, only vignette data will be collected and fed back to providers. Feedback will consist of specific data on vignette outcome scores for the individual physicians and for the sites overall.
2. Site Selection: Primary care clinics at 2 VAMCs
3. Study Population and Sampling: We will enroll primary care physicians at 2 VAMCs. 30 consenting physicians will be prospectively randomized into two groups. One group will receive feedback of their vignette scores, and the other group will serve as control, receiving no feedback.
4. Variables and Measurement Instruments: Computerized vignettes measuring clinical practice completed by the physicians for diabetes, CAD, COPD, and Depression and a composite health outcome measures from the medical records of these physicians� patients with diabetes and CAD.
5. Data Collection Strategy and Timeline: Vignettes will be administered to all physicians at baseline, with feedback of scores 3 months later and readministration of vignettes 9 months thereafter to measure the trend in improvement. The composite outcome data will only be collected at baseline only.
6. Data Analysis: The statistical analysis will compare the effects within the context of an analysis of covariance (ANCOVA) model. The analyte is the quality of care physicians give to patients with four common conditions. The relationship between vignette scores and patient outcomes will be modeled accounting for clustering effects. The prospective experimental design will be used to quantify possible differences between the intervention and control groups. The data will be analyzed using a three-way crossed, one-way nested ANCOVA model where the covariate is the baseline vignette score. This model can be used to look at case effects, by domain, level of training, and by site.

ELIGIBILITY:
Inclusion Criteria:

Physician at SF VAMC with panel of primary care patients

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-09; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Disease-specific patient care indicators, comparing results at six months.

CONTACTS AND LOCATIONS:
Overall Officials: Sharad Jain, MD, Principal Investigator — San Francisco
Locations (1):
- San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Peabody JW, Luck J, Jain S, Bertenthal D, Glassman P. Assessing the accuracy of administrative data in health information systems. Med Care. 2004 Nov;42(11):1066-72. doi: 10.1097/00005650-200411000-00005. PMID 15586833